CLINICAL TRIAL: NCT02590159
Title: Clinical Study for the BONGO NASAL EPAP Device in the Treatment of Obstructive Sleep Apnea (OSA)
Brief Title: Clinical Study for the BONGO NASAL Expiratory Positive Airway Pressure (EPAP) Device in the Treatment of Obstructive Sleep Apnea (OSA)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: delay in enrollment
Sponsor: InnoMed Healthscience Inc. (Industry)
Collaborators: RVW Clinical Consulting (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INN-C002
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: BONGO NASAL EPAP — The BONGO NASAL EPAP device consists of two nasal inserts (a connected pair), each containing an actuated valve, with a patient attachment mechanism. The device works by providing an inhalation port that offers minimal inhale resistance during inhalation, but is closed by the actuated valve so that exhalation occurs against a fixed orifice. This mechanism provides increased EPAP upon exhalation.

SUMMARY:
Single center clinical study for the BONGO NASAL EPAP device in the treatment of obstructive sleep apnea for the purpose of obtaining safety and efficacy data

ELIGIBILITY:
Inclusion Criteria:

* Capacity and willingness to sign informed consent
* ≥ 21 years of age
* Diagnosis of mild to moderate OSA (AHI ≥ 5 and AHI < 30) within 12 months of the screening visit.
* Able to tolerate using the device during a day time trial/acclimation
* Are currently using CPAP or have been prescribed CPAP and are considered CPAP non-adherent (as per either their CPAP data card and/or verbal confirmation of a diagnosis and unwillingness to use CPAP)

Exclusion Criteria:

* Nasal deformities
* Severe nasal allergies
* Rhinitis or moderate nasal congestion, acute upper respiratory (including nasal, sinus or middle ear) inflammation or infection, or perforation of the ear drum
* Co-morbid sleep disorders
* Currently on a hypnotic for insomnia (who have had insomnia for more than a month and take a hypnotic on a daily basis and/or transient insomnia being treated)
* Uncontrolled or serious illness, including but not limited to: severe breathing disorders including hypercapnic respiratory failure, respiratory muscle weakness, bullous lung disease (as seen in some types of emphysema), bypassed upper airway, pneumothorax, pneumomediastinum, etc.; severe heart disease (including heart failure); or pathologically low blood pressure.
* Full Face Mask user
* Mouth breather
* Pregnant (Female subjects of child bearing age will be asked if they are and/or planning on becoming pregnant during the study; acceptable methods of birth control include birth control pills and barrier method)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Lamaie, MD, Principal Investigator — Sleep Therapy and Research Center
Locations (1):
- Sleep Therapy and Research Center, San Antonio, Texas, United States